CLINICAL TRIAL: NCT04956328
Title: A Multi-center, Randomized, Double-blind Trail Evaluating the Efficacy and Safety of Combination of Obecholic Acid and UDCA Compared With UDCA Monotherapy in PBC Patients With an Inadequate Response to UDCA .
Brief Title: Study of Obeticholic Acid（OCA） Combination With Ursodeoxycholic Acid (UDCA) in Patients With Primay Biliary Cirrhosis (PBC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABDS-CS-01
Record Dates: First submitted 2021-07-01; First posted 2021-07-09 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCA Tablets 5-10 mg (Experimental): OCA 5 mg once daily in combination with UDCA for 24 weeks and then titrating up to 10 mg based on tolerability and response for remainder of double-blind period.
  Interventions: Drug: Obeticholic Acid Tablets; Drug: UDCA
- Placebo (Placebo Comparator): Placebo once daily in combination with UDCA for 48 weeks.
  Interventions: Drug: UDCA; Drug: Placebo

INTERVENTIONS:
Drug: Obeticholic Acid Tablets — Obeticholic Acid：Once a day (QD) by mouth (PO).
  Arms: OCA Tablets 5-10 mg
Drug: UDCA — UDCA：continue prestudy dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Obecholic acid is a modified bile acid and Farnesoid X receptor (FXR) agonist. FXR is a key regulator of bile acid synthesis and transport. Bile acids are used by the body to help with digestion. Conventional therapy with obecholic acid will improve liver function of patients with PBC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 75 years.
2. Meet at least 2 of the following 3 PBC diagnoses:

   1. Patients had elevated alkaline phosphatase for at least 3 months before enrolment.
   2. AMA positive (titer ≥1:40), or if AMA negative, PBC specific antibodies (anti- GP210 and/or anti-SP100 and/or AMA-M2) are required.
   3. Liver biopsy suggested PBC 48 weeks before enrollment.
3. ALP > 1.67× ULN before enrollment.
4. Taking UDCA with stable dose for at least 3 months before enrollment.

Exclusion Criteria:

1. Merging with other virus infected.
2. With other existing liver disease or a history of liver disease.
3. With clinical complications of PBC or clinically significant hepatic decompensation.
4. Child-pugh grade B or C.
5. Creatinine (Cr) ≥ 1.5×ULN and serum creatinine clearance rate < 60mL/min; [Calculation formula: Cr:(140-age)×weight(kg) /0.818 × Scr (μmol/L)，female Cr=Cr × 0.85].
6. ALT or AST>5×ULN;Tbil > 2×ULN.
7. Patients with a history of severe pruritus 2 months before enrollment.
8. The presence of clinically relevant arrhythmias or associated history that may affect survival during the study period.
9. With diseases that may cause nonhepatic ALP increases (e.g., Paget's disease) or which may diminish life expectancy to < 2 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of PBC patients reaching the compound endpoint after 48 weeks of treatment (Compound endpoint: alkaline phosphatase (ALP) < 1.67× Upper Limit of Normal(ULN), ALP decrease by at least 15% , and total bilirubin ≤ ULN ) | up to 48 weeks
  Compound endpoint: ALP < 1.67× ULN, ALP decrease by at least 15% , and total bilirubin ≤ ULN

SECONDARY OUTCOMES:
Percentage of PBC patients reaching the compound endpoint after 4 weeks, 12 weeks, 24 weeks and 36 weeks of treatment (Compound endpoint: ALP < 1.67× ULN, ALP decrease by at least 15% , and total bilirubin ≤ ULN ) | up to 36 weeks
  Compound endpoint: ALP < 1.67× ULN, ALP decrease by at least 15% , and total bilirubin ≤ ULN
Rate of change of liver function indicators from baseline | up to 48 weeks
  Liver function: ALP (alkaline phosphatase ), ALT (Alaninetransaminase), AST(aspartate transaminase), GGT( γ-glutamyl transpeptadase ), TBA (total bile acid) and Tbil (total bilirubin)

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China